CLINICAL TRIAL: NCT00614419
Title: Prospective Randomized, Double-blind, Controlled Trial Comparing Lichtenstein's Repair of Inguinal Hernia With Polypropylene Mesh Versus Surgisis ES Soft Tissue Graft
Brief Title: Prospective Randomized Trial Comparing Lichtenstein's Repair of Inguinal Hernia With Polypropylene Mesh Versus Surgisis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Dr. Luca Ansaloni, Unit of Surgery, St.Orsola-Malpighi Hospital - University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81/2002/O
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Hernia, Inguinal
Keywords: Hernioplasty; polypropylene; extracellular matrix; xenograft
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The Lichtenstein tension-free hernioplasty with polypropylene mesh
  Interventions: Device: Prolene Polypropylene Mesh
- 2 (Experimental): The Surgisis mesh group: in this group of patients a 7x20cm Surgisis ES Soft Tissue Graft sheet will be used. In sterile manner the sheet will be removed from the peel-open package. The Surgisis sheet will be cut and fashioned as appropriate. Then the pre-shaped sheet will will be placed for at least 10 minutes into a sterile dish with sterile room-temperature normo-saline to be rehydrated. Using aseptic techique, the rehydrated Surgisis sheet will be transferred to the already prepared and dissected inguinal region and will be fixed with PDS II 2/0.
  Interventions: Device: Surgisis Inguinal Hernia Matrix

INTERVENTIONS:
Device: Prolene Polypropylene Mesh — The Lichtenstein tension-free hernioplasty consists of a swatch of polypropylene mesh, partway slit 1 cm from its inferior edge to accommodate the spermatic cord. The mesh is sutured circumferentially to the internal oblique abdominal muscle, the rectus sheath and the shelving edge of the inguinal ligament. The tails of the mesh are drawn around the cord and the inferior edge of each tail is sutured to the inguinal ligament. In case of direct hernias, no effort is made to repair the hernia itself. In indirect hernias the sac is excised, except for sliding hernias. The polypropylene mesh group: in this group of patients the polypropylene mesh will be fixed by the above mentioned sutures in Prolene 3/0.
  Other Names: PP
  Arms: 1
Device: Surgisis Inguinal Hernia Matrix — The Surgisis mesh group: in this group of patients a 7x20cm Surgisis ES Soft Tissue Graft sheet will be used. In sterile manner the sheet will be removed from the peel-open package. The Surgisis sheet will be cut and fashioned as appropriate. Then the pre-shaped sheet will will be placed for at least 10 minutes into a sterile dish with sterile room-temperature normo-saline to be rehydrated. Using aseptic techique, the rehydrated Surgisis sheet will be transferred to the already prepared and dissected inguinal region and will be fixed with PDS II 2/0.
  Other Names: SIHM
  Arms: 2

SUMMARY:
To evaluate the safety and efficacy of the Lichtenstein's hernioplasty using the Surgisis ES soft tissue graft, as a mesh, and to compare it with the traditional Lichtenstein procedure performed with polypropylene mesh.

DETAILED DESCRIPTION:
Inclusion and Exclusion Criteria

Inclusion criteria:

* Male, adult patients
* ASA I-III patients
* Non-complicated primary inguinal hernia (classification according to Gilbert I-II-III-IV-V-VI, modified. according to Rutkow and Robbins) performed in non-emergency setting and repaired with a Lichtenstein's hernioplasty using polypropylene or Surgisis mesh
* Informed consent

Exclusion criteria

* Recurrent hernias
* Any condition preventing a correct evaluation of pain (non-cooperative patient, blind patient, drug addicted)
* Hypersensitivity to any drug in study
* Patients with an intra-operative findings of different pathology will be excluded from the study

Outcomes:

General objectives of the study will be:

1. to determine the safety of the Lichtenstein's hernioplasty with Surgisis ES by noting any complications observed intraoperatively and postoperatively
2. to determine the efficacy of the Lichtenstein's hernioplasty with Surgisis ES in comparison with the traditional method with polypropylene mesh by noting the grade of postoperative pain, discomfort, quality of life, the rate of wound infection and other complications, and the recurrence rate.

The specific objectives of the study will be:

1. to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), simple verbal scale (SVS) and parenteral/oral analgesic consumption in the two groups.
2. to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS) and simple verbal scale (SVS).
3. to measure the postoperative health general status and quality of life with the Short Form 36 (SF-36) questionnaire.
4. to rate the wound infection risk.
5. to monitor any other postoperative complication observed in the immediate, mid-term and long-term postoperative period.
6. to measure the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Male, adult patients
* ASA I-III patients
* Non-complicated primary inguinal hernia (classification according to Gilbert I-II-III-IV-V-VI, modified. according to Rutkow and Robbins) performed in non-emergency setting and repaired with a Lichtenstein's hernioplasty using polypropylene or Surgisis mesh
* Informed consent

Exclusion Criteria:

* Recurrent hernias
* Any condition preventing a correct evaluation of pain (non-cooperative patient, blind patient, drug addicted)
* Hypersensitivity to any drug in study
* Patients with an intra-operative findings of different pathology will be excluded from the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), simple verbal scale (SVS) and parenteral/oral analgesic consumption in the two groups | 1 week, 1, 3, 6 months, 1, 2, 3, 4, 5 years

SECONDARY OUTCOMES:
to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS) and simple verbal scale (SVS). | 3, 6 months, 1, 2, 3, 4, 5 years
to rate the wound infection risk. | 1 week, 1, 3, 6 months, 1, 2, 3, 4, 5 years
to monitor any other postoperative complication observed in the immediate, mid-term and long-term postoperative period. | 1 week, 1, 3, 6 months, 1, 2, 3, 4, 5 years
to measure the recurrence rate | 1 week, 1, 3, 6 months, 1, 2, 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ansaloni, MD, Principal Investigator — St.Orsola-malpighi Hospital
Locations (1):
- St.Orsola-Malpighi University Hospital, Bologna, Italy